CLINICAL TRIAL: NCT06950086
Title: A Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of the CDK2/4/6 Inhibitor TYK-00540 Tablets in Patients With Advanced Solid Tumors
Brief Title: Study of TYK-00540 Tablets in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYKM5807101
Record Dates: First submitted 2025-04-11; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: HR-positive, HER2-negative Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TYK-00540±Fulvestrant (Experimental): TYK-00540• Find the maximum tolerated dose(MTD) and the recommended phase 2 dose (RP2D) of TYK-00540, given orally. • Increased dose cohorts from low dose to MTD, starting at 5mg twicely.
  fulvestrant: is in the form of a syringe containing 5ml of an injection solution of 250mg of fulvestrant for injection. The recommended dose is every 28 days, once at a dose of 500mg, and on the 15th day after the initial injection, a loading dose of fulvestrant 500mg id added.
  Interventions: Drug: TYK-00540

INTERVENTIONS:
Drug: TYK-00540 — Increased dose cohorts from low to MTD (5mg Cohort 1;10 mg Cohort 2; 20 mg Cohort 3; 30 mg Cohort 4;40 mg Cohort 5) decreased dose cohorts for the combination (TYK-00540 30 mg+Fulvestrant Cohort 1;TYK-00540 20mg +Fulvestrant)

SUMMARY:
This study is to evaluate the safety, pharmacokinetics, and preliminary antitumor activity of TYK-00540 as monotherapy or combined with fulvestrant in advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multi-center, dose-escalation and expansion phase I/II study to evaluate dose limiting toxicities (DLT) and determine the maximum tolerated dose (MTD) in subjects with locally advanced or metastatic solid tumors.

To investigate the pharmacokinetic profile of TYK-00540 and its metabolites after single then multiple doses of TYK-00540 administered orally once daily. To assess preliminary effectiveness. To evaluate the efficacy of TYK-00540 combined with fulvestrant in subjects with ER+/HER2- breast cancer who have relapsed or progressed after treatment with CDK4/6 inhibitors

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, gender requirements:

   Monotherapy dose-escalation phase: No gender restriction.

   Combination dose-selection phase: No gender restriction.

   Monotherapy and combination expansion phases:

   Cohort A-1: Females only.

   Other cohorts: No gender restriction.

   Monotherapy Dose-Escalation Phase:
2. Histologically or cytologically confirmed locally advanced/metastatic solid tumors with no standard treatment available, failure of/intolerance to standard treatment, or refusal of standard treatment.

   Monotherapy Dose-Expansion Phase:

   Cohort A-1: Histologically or cytologically confirmed advanced platinum-resistant epithelial ovarian cancer (EOC)/fallopian tube cancer/primary peritoneal cancer:

   Platinum resistance defined as: Disease recurrence/progression <6 months after completion of prior platinum-based chemotherapy (≥4 cycles) or progression during initial/recurrent treatment.

   Disease recurrence/progression requires:
   1. Objective radiographic progression; OR
   2. Persistent CA125 elevation (confirmed after 1 week) with clinical symptoms or signs of progression.

      * 3 prior lines of chemotherapy for recurrent/metastatic disease, with ≤1 systemic therapy after platinum resistance.

   Cohort A-2: HR+/HER2- advanced breast cancer with confirmed resistance to CDK4/6 inhibitors (≥1 documented instance).

   Combination Dose-Selection Phase:

   HR+/HER2- advanced breast cancer with confirmed resistance to CDK4/6 inhibitors (≥1 documented instance).

   Combination Dose-Expansion Phase:

   Cohort B-1: HR+/HER2- advanced breast cancer with prior endocrine therapy resistance and either:

   No prior CDK4/6 inhibitor treatment; OR

   CDK4/6 inhibitor-treated in the adjuvant setting with recurrence >1 year after completion (no confirmed resistance).

   Cohort B-2: HR+/HER2- advanced breast cancer with progression during/after endocrine + CDK4/6 inhibitor therapy:

   For adjuvant CDK4/6 inhibitor resistance: Recurrence during or ≤1 year after treatment;

   ≥1 documented CDK4/6 inhibitor resistance.

   Note for Cohorts A-2, Combination Dose-Selection, and Combination Expansion Phases:
   * 2 prior endocrine therapy regimens for recurrent/metastatic disease (adjuvant endocrine therapy leading to recurrence within 1 month of completion counts as 1 regimen).
   * 1 prior chemotherapy or ADC regimen for recurrent/metastatic disease.

   Prior CDK4/6 inhibitor use:
   1. Duration ≥6 months;
   2. Adjuvant CDK4/6 inhibitor use with progression >1 year after completion does not count as resistance;
   3. Switching CDK4/6 inhibitors due to intolerance is permitted.
3. For female patients in Combination Phases:

   Meet ≥1 of the following:
   1. Bilateral oophorectomy;
   2. Age ≥60 years;
   3. Age <60 years with natural menopause ≥12 months (without chemotherapy, tamoxifen, toremifene, or ovarian suppression in the past year), confirmed by postmenopausal FSH and estradiol levels;
   4. Age <60 years on tamoxifen/toremifene with postmenopausal FSH and estradiol levels.

   Non-postmenopausal patients must use LHRH agonists/antagonists throughout the study.
4. Baseline Lesions:

   Monotherapy dose-escalation: Extracranial evaluable/measurable lesions.

   Combination phases: Extracranial measurable lesions (RECIST 1.1).
5. ECOG performance status 0-1, no deterioration within 2 weeks prior to first dose (Appendix II).
6. Life expectancy ≥3 months.
7. Adequate Organ Function:

   Liver:TBIL ≤1.5×ULN, ALT/AST ≤2.5×ULN (≤5×ULN for liver metastases; ≤3×ULN for combination with fulvestrant).

   Kidney:Serum creatinine ≤1.5×ULN, creatinine clearance ≥50 mL/min (Cockcroft-Gault formula, Appendix III).

   Hematology:Platelets ≥90×10^9/L, ANC ≥1.5×10^9/L, Hb ≥90 g/L (without transfusion/G-CSF within 2 weeks).

   Cardiac:LVEF ≥50% (echocardiogram), QTcF <470 ms. Coagulation:INR ≤1.5, APTT ≤1.5×ULN (without anticoagulation).
8. Contraception:Females of childbearing potential: Negative pregnancy test and commitment to highly effective contraception/abstinence from screening until 6 months post-treatment (Appendix IV).Males: Commitment to contraception/abstinence during the same period.For fulvestrant combination: Contraception until 1 year after last dose.
9. Voluntary signed ICF (or by legal guardian) and willingness to comply with study procedures.

Exclusion Criteria:

1. Known hypersensitivity to any excipient of TYK-00540 or contraindication to fulvestrant (for Combination Dose-Selection and Combination Expansion Phases).
2. Prior/concurrent therapies:

   Systemic anticancer therapies within 28 days prior to first dose: chemotherapy, large-molecule targeted therapy, immunotherapy.

   Endocrine therapy, small-molecule targeted therapy, or fluorouracil-based oral agents within 14 days prior to first dose.

   Nitrosoureas or mitomycin within 6 weeks prior to first dose. Anticancer herbal medicine or traditional Chinese medicine within 7 days prior to first dose.

   Local radiotherapy (e.g., thoracic/rib) or palliative radiotherapy for bone metastases within 7 days prior to first dose.

   Major surgery (excluding minor procedures, e.g., appendectomy, tumor biopsy) within 4 weeks prior to first dose.

   Proton pump inhibitor (PPI) use within 7 days prior to first dose or during the study.

   Concurrent use of medications known to prolong QTc interval or induce torsades de pointes (Appendix V).

   Participation in other interventional clinical trials within 28 days prior to first dose (non-interventional trials excluded).

   Prior allogeneic bone marrow transplantation. For Combination Phases: prior use of fulvestrant, other SERDs, or SERCAs.
3. History of other malignancies, except:Cured basal cell carcinoma, squamous cell carcinoma, cervical carcinoma in situ, thyroid papillary carcinoma, ductal carcinoma in situ of the breast, or malignancies with disease-free survival >3 years.
4. Residual toxicity from prior therapy >Grade 1 (except alopecia or platinum-related neuropathy).
5. Central nervous system (CNS) disease:Primary CNS tumors, CNS metastases with prior local treatment failure, or newly diagnosed CNS metastases.Exception: Asymptomatic, stable CNS metastases (no steroids/CNS-specific treatment ≥14 days, radiologically confirmed stability at screening).
6. Spinal cord compression caused by tumor.
7. Visceral crisis.
8. Clinically uncontrolled pleural effusion, ascites, or pericardial effusion requiring repeated drainage/medical intervention (within 14 days prior to first dose).
9. Clinically significant ECG abnormalities at baseline (e.g., QTc ≥470 ms, complete LBBB, acute/indeterminate-age myocardial infarction, ST-T changes suggesting ischemia, second-/third-degree AV block, severe bradycardia/tachycardia).
10. Cardiovascular events within 6 months:Myocardial infarction, long QT syndrome, torsades de pointes, arrhythmias (sustained ventricular tachycardia/fibrillation), severe conduction defects (e.g., bifascicular block, third-degree AV block), unstable angina, coronary/peripheral bypass, symptomatic CHF (NYHA Class III/IV), stroke, TIA, symptomatic pulmonary embolism, or clinically significant thromboembolism.Persistent NCI CTCAE ≥Grade 2 arrhythmia, atrial fibrillation (asymptomatic atrial fibrillation ≥Grade 2).

    Exception: Patients with cardiac pacemakers/devices and QTcF >470 ms may be eligible after discussion with the medical monitor.
11. Unstable or uncontrolled medical conditions affecting safety/compliance, including:Uncontrolled hypertension (systolic BP >160 mmHg and/or diastolic BP >100 mmHg).Uncontrolled diabetes, active bleeding, ocular disease, severe psychiatric/neurological/cardiovascular/respiratory disorders.
12. Active/uncontrolled infections or immunodeficiencies:Active HBV (HBsAg-positive with HBV DNA ≥2000 copies/mL [or 500 IU/mL]).Active HCV (HCV antibody-positive with HCV RNA-positive).HIV-positive.Exception: Asymptomatic chronic HBV/HCV carriers.
13. Lung disease:Radiation pneumonitis requiring steroids, interstitial lung disease (ILD)/pneumonitis (active or drug-induced), acute/progressive pulmonary fibrosis, or high-risk factors for ILD per investigator judgment.
14. Clinically significant gastrointestinal disorders affecting drug absorption (e.g., dysphagia, uncontrolled vomiting, active ulcers, inflammatory bowel disease, chronic diarrhea, bowel obstruction, chronic PPI-dependent conditions).
15. Hypercoagulability with thromboembolic events within 6 months (e.g., stroke, DVT, pulmonary embolism).
16. Pregnancy, lactation.
17. The investigator concluded that the patient was not suitable to participate in the study (such as not conforming to the most beneficial treatment for the patient, patient compliance, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Within 31 days of the first dose
  Numbers of participants experiencing AEs which are defined as DLTs classfied by CTCAE
Recommended dose for combination-agent escalation and single-agent expansion (RDE) | 1 year
  To determine the recommended dose for combination-agent escalation and single-agent expansion agent expansion.
Adverse events (AEs) | From Baseline up to 28 days after the end of the treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Objective response rate (ORR) | At least 24 weeks
  ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

SECONDARY OUTCOMES:
The time to the peak concentration (Tmax) | 0 hours (h) (within 30 min before dosing), 0.25 h, 0.5 h , 1 h , 2 h , 3 h, 4 h, 8 h , 12 h, 24 h after dosing
  Tmax is defined as the time of maximum concentration of the drug in blood observed after a drug dose administration.
Maximum plasma concentration (Cmax) | 0 hours (h) (within 30 min before dosing), 0.25 h, 0.5 h , 1 h , 2 h , 3 h, 4 h, 8 h , 12 h, 24 h after dosing
  Cmax is the maximum (or peak) plasma concentration that the drug achieves in blood after the drug has been administered.
Minimum plasma concentration (Cmin) | 0 hours (h) (within 30 min before dosing), 0.25 h, 0.5 h , 1 h , 2 h , 3 h, 4 h, 8 h , 12 h, 24 h after dosing
  Cmin is the minimum plasma concentration that the drug achieves in blood after the drug has been administered.
Disease Control Rate (DCR) | At least 24 weeks
  DCR is defined as the proportion of patients with a best overall response of complete response (CR) , partial response (PR) or Stable disease (SD) ≥6 weeks during the study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No